Official Title: LCI-HEM-PCNSL-RMPV-001: A Phase 1B Trial Nivolumab Consolidation Following Completion of High-Dose Methotrexate Containing Induction Chemotherapy in Older (≥ 65) Patients With Primary CNS Lymphoma NCT04022980

IRB-Approved Date: 08/25/2022

# ATRIUM HEALTH CONSENT TO PARTICIPATE IN A RESEARCH STUDY

Sponsor / Study Title: Levine Cancer Institute / A Phase 1B Trial of Nivolumab

Consolidation Following Completion of High-Dose

Methotrexate Containing Induction Chemotherapy in Older (≥

65) Patients with Primary CNS Lymphoma

Protocol Number: LCI-HEM-PCNSL-RMPV-001

Principal Investigator:

(Study Doctor)

Steven Park, MD

Telephone: (24 Hours) (24 Hours)

Address: Levine Cancer Institute - Carolinas Medical Center

Please read this form carefully. Take time to ask the study doctor or study staff as many questions about the study as you would like. The study doctor or study staff can explain words or information that you do not understand. Reading this form and talking to the study doctor or study staff may help you decide whether to take part or not. If you decide to take part in this study, you must sign and date your name at the end of this form. You cannot take part in this research study until you sign and date this form.

This form is for use in a research study that may involve subjects who may or may not have the capacity to consent to take part in the study. Accordingly, when the subject cannot legally consent to take part, pronouns "you" and "your" should be read as referring to the subject rather than the person (legally authorized representative) who is signing this form for the subject.

#### INTRODUCTION TO THE RESEARCH STUDY

The Study Doctor listed on the first page of this form is asking you to participate in this research study at Levine Cancer Institute (LCI) and Atrium Health to evaluate the safety and efficacy (how well it works) of the study treatment, nivolumab given after completion of a high dose methotrexate containing chemotherapy induction regimen in subjects 65 years or older with primary CNS (central nervous system) lymphoma (PCNSL).

Steven Park, MD

Advarra IRB Approved Version 25 Aug 2022

Revised 25 Aug 2022



Affix Participant Barcode Label Here

You are being asked to take part in this study because you have primary CNS lymphoma previously treated with a high-dose methotrexate containing chemotherapy (called "induction"), are 65 years or older, and are not eligible for whole brain radiation therapy or ASCT (autologous stem cell transplant - where your normal blood stem cells are given back to you after high dose chemotherapy).

This is a clinical trial, a type of research study. Your study doctor will explain the clinical trial to you. Clinical trials include only people who choose to take part. Please take your time to decide on study participation. You have also been told that you have the option not to participate. You may discuss your decision with your friends and family. You can also discuss it with your healthcare team. If you have any question, you can ask your study doctor for more explanation.

This study is being carried out under the sponsorship of Levine Cancer Institute (LCI). Bristol-Myers Squibb (BMS) is the company that makes the study drug nivolumab and will be providing it in this study. Nivolumab is currently approved by the FDA (Food and Drug Administration) for relapsed or progressed Hodgkin lymphoma (HL) but is not FDA approved for your condition and is therefore considered experimental.

Taking part in this study is entirely voluntary.

#### PURPOSE OF THE RESEARCH STUDY

Research studies are done to find out the best way to treat patients.

Primary central nervous system (CNS) lymphoma is a disease in which malignant (cancer) cells form in the lymph tissue of the brain and/or spinal cord and sometimes in the eyes. Approximately 25% of patients with PCNSL do not respond to first line therapy and more than 50% relapse (disease returns) and these numbers worsen in older patients with PCNSL. Therefore, new approaches to treatment are urgently needed, especially for older PCNSL patients.

The study drug, nivolumab, is an antibody (a type of human protein) that is being evaluated to see if it will stimulate the body's immune system to work against tumor cells. Nivolumab has been clinically shown to be effective in a small study of PCNSL. Treatment with a high-dose methotrexate (HD-MTX) containing induction chemotherapy regimen (such as the combination of rituximab, methotrexate, procarbazine, vincristine [R-MPV]) is one of the most commonly used chemotherapy treatments in PCNSL. This study will evaluate the safety of treatment with nivolumab after HD-MTX containing induction chemotherapy. Another study goal is to evaluate how effective treatment with nivolumab given after completion of HD-MTX containing induction chemotherapy is in treating PCNSL.

### HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

You will be one of approximately 20 subjects to participate in this study at approximately 2-4 participating sites.

Steven Park, MD


Revised 25 Aug 2022

Affix Participant Barcode Label Here

#### **HOW THE STUDY WORKS**

This study will include 2 stages:

Stage 1 will include up to 6 subjects to determine the safety of nivolumab after completion of HD-MTX containing induction chemotherapy.

Stage 2 will include up to 14 subjects to learn how effective nivolumab is after completion of HD-MTX containing induction chemotherapy.

It is expected that you will have around 6 months of study treatment and then 3-5 years of follow-up while on this study.

Before the study starts, you will be asked to sign and date this consent form. If you agree to participate in the study and sign and date the consent form, the study doctor will do some tests and procedures to find out if you can be in the study.

## Before you begin the study (Baseline):

- Medical and disease history
- Physical exam, weight and performance status (scale used to assess how active you are)
- Vital signs (temperature, blood pressure, and heart rate)
- You will be asked how you are feeling, and any symptoms you might have before you start study treatment will be documented.
- You will be asked about any medication you use (prescription, over the counter, supplements).
- HBV DNA testing (tests for exposure to the hepatitis B virus) The study doctor may be required by law to report the result of this test to the local health authority.
- Neurologic Assessment in Neuro-Oncology (NANO) assessment (evaluates brain and nervous system function)
- Radiologic tests:
  - O MRI (Magnetic Resonance Imaging) is a technique that uses a magnetic field and radio waves to create detailed images of the organs and tissues within your brain or spine.
- Laboratory assessments:
  - o Complete Blood Count with Differential (CBCD evaluates the cells that circulate in blood)
  - Comprehensive Metabolic Panel (CMP gives a snapshot of the body's blood chemistry)
  - o Lactate Dehydrogenase (LDH checks for tissue damage in the body)
  - O Thyroid Stimulating Hormone (TSH), Thyroxine (T4), free triiodothyronine (T3) (measures thyroid gland function)

Steven Park, MD


- Serum (blood) or urine pregnancy test for women of childbearing potential
- Collection of archival tumor tissue (previously collected, stored tumor samples)
- If a lumbar puncture (spinal tap taking a sample of the liquid that fills and surrounds the brain and the spinal cord) is being performed to check for disease involvement in your cerebrospinal fluid during the screening period, a portion of the cerebrospinal fluid sample will be collected for correlative studies.

  Correlative studies look at the relationship between drugs and the effects they have on the body.

Many of these tests may be repeated during the course of this research study.

If you are having unfavorable side effects, the study treatment may be stopped for a while, or the dose of the study drug(s) may be reduced. Your study doctor will also discuss with you whether it is in your best interest to continue the study treatment. You will continue study treatment until completion or until study treatment is interrupted for any reason.

# Description of all visits, including timing of visits:

Nivolumab will be given IV over 30 minutes on Day 1 of 28-day cycles for up to 6 cycles.

# Day 1 Nivolumab (plus or minus 2 days)

- Medical history, physical examination, weight and performance status (scale used to assess how active you are)
- Vital signs
- Laboratory assessments:
  - o CBCD
  - o CMP
  - o LDH
  - o TSH, free T4, T3 (Day 1 of Cycle 1 and Cycle 4 only)
  - o Serum or urine pregnancy test for women of childbearing potential (within 3 days prior to the first dose of nivolumab and then D1 of every cycle)
- You will be asked about any medication you use (prescription, over the counter, supplements).
- You will be asked how you are feeling, and any symptoms (side effects) you are experiencing will be documented.

Steven Park, MD


# After Cycle 3 Nivolumab (14 plus or minus 7 days)

- Radiologic assessments: MRI of brain and/or spine.
- Informed Consent: If your disease has progressed, your study doctor recommends that you continue study treatment with nivolumab and you wish to continue to receive study treatment with nivolumab, you will be asked to sign and date a separate consent form.

# After Nivolumab Study Treatment (8 plus or minus 2 weeks after the last cycle of Nivolumab)

- Medical history, physical examination, weight and performance status
- Vital signs
- NANO assessment
- Laboratory assessments:
  - CBCD
  - o CMP
  - o LDH
  - o TSH, free T4, T3
- You will be asked about any medication you use (prescription, over the counter, supplements).
- You will be asked how you are feeling, and any symptoms (side effects) you are experiencing will be documented.
- Radiologic assessments: MRI of brain and/or spine.
- Lumbar puncture may be performed to collect a sample of CSF (cerebrospinal fluid) to evaluate your disease and for correlative studies only if previous lumbar punctures showed evidence of disease in your cerebral spinal fluid.

# Follow-Up

Active follow-up including radiologic assessments will occur approximately every 4 months for 1 year, then every 6 months for 1 year and then at the frequency as determined by your study doctor until the study has been completed. Active follow-up will continue until your disease worsens or you start new cancer treatment. If your disease progresses during nivolumab study treatment, you will be contacted by phone approximately every 6 months to see how you are doing. If we are unable to reach you by phone, we will attempt to contact you by mail.

Active follow-up Visit procedures (if your disease does not progress during nivolumab study treatment):

- Medical history, physical examination, weight and performance status
- Vital signs
- NANO assessment

Steven Park, MD


- Laboratory assessments:
  - o TSH, free T4, T3
- Radiologic assessments: MRI of brain and/or spine

#### YOUR ROLE IN THE STUDY

Taking part in a research study can be an inconvenience to your daily life. Please consider the study time commitments and responsibilities as a research subject when you are deciding to take part. Your responsibilities as a study subject include the following:

- Tell the truth about your medical history and current conditions.
- Tell the study doctor if you have been in a research study in the last 30 days or are in another research study now.
- Tell the study doctor about any problems you have during the study.
- The study doctor or study staff will talk to you about any food or medicines that you should not take while in this study.

#### RISKS OF THE STUDY

As with all research studies, the study drugs and study procedures may involve unknown risks. Any medication can have temporary or permanent side effects and can cause unforeseen adverse reactions.

You may have side effects while on the study. Everyone taking part in the study will be monitored carefully for any side effects. Side effects may be mild or very serious. Your study doctor may give you medicines to help lessen side effects. Many side effects go away soon after you stop taking the study drug. In some cases, side effects can be serious, long lasting, or may never go away.

Any drug has risks and side effects which may vary from person to person. Side effects may be mild or very severe. Side effects seen on research studies can result from a subject's disease, the drug under study, other drugs you are taking, other diseases you have, or a combination of these.

#### Nivolumab Risks

Nivolumab may cause one or more of the side effects listed below. This information is based on data from cancer subjects in other clinical trials with nivolumab. In addition, there may be side effects that are not yet known that may occur. These may be life threatening or lead to death. You should tell the study staff right away about any possible side effects you experience.

Steven Park, MD


Very common side effects of nivolumab are [greater than or equal to 1/10 or greater than or equal to 10%]:

- Diarrhea
- Feeling tired or lack of energy
- Skin itching
- Skin rash

Common side effects of nivolumab include [greater than or equal to 1/100 to less than 1/10 or greater than or equal to 1% to less than 10%]:

- Abdominal (belly) pain
- Alkaline phosphate increased: lab test result associated with liver or bone abnormalities
- Allergic reaction/hypersensitivity, a reaction related to infusion of the study drug. The symptoms may include but not limited to fever, rash, pain, swelling.
- ALT increased: lab test result associated with abnormal liver function
- Amylase increased: lab test result associated with pancreas inflammation
- AST increased: lab test result associated with abnormal liver function
- Bilirubin increased, lab test associated with abnormal liver function
- Chills
- Constipation
- Cough
- Creatinine increased: lab test result associated with decreased kidney function
- Decreased appetite
- Dizziness or vertigo (feeling off balance which can lead to dizziness)
- Dry mouth
- Dry skin
- Fever
- Headache
- High blood pressure
- Increased blood sugar, a lab test result or diabetes, a disease that results in too much sugar in the blood
- Inflammation of the colon.
- Inflammation of the mouth
- Lipase increased: lab test result associated with pancreas inflammation
- Loss of color (pigment) from areas of skin
- Low sodium levels in the blood
- Low platelet counts (thrombocytopenia): this may increase your risk for skin bruising, nose bleeds, and bleeding from the gums
- Low red blood cell counts (anemia), this may make you feel weak and tired

Steven Park, MD


- Lung inflammation (pneumonitis): Inflammation of the tissues of the lung. While many subjects with x-ray or CT abnormalities have not developed any symptoms, some subjects have developed mild to severe symptoms of their lung inflammation. Signs and symptoms of lung inflammation may include difficulty breathing, pain or discomfort while breathing, chest pain, cough, shortness of breath, increased rate of breathing, fever, low blood oxygen levels, or fatigue.
- Nausea
- Pain in the muscles, bones, ligaments, tendons and nerves
- Shortness of breath
- Swelling, including face, arms, and legs (edema)
- Thyroid gland function decreased or may be increased, thyroid stimulating hormone a lab test result associated with abnormal thyroid function
- Tingling, burning, numbness or weakness, possibly in arms, legs, hands and feet
- Vomiting

# <u>Uncommon side effects of nivolumab include [greater than or equal to 1/1,000 to less than 1/100 or greater than or equal to 0.1% to less than 1%]:</u>

- A common viral / bacterial infection that affects the nose, throat, and airways (upper respiratory tract infection)
- A condition in which not enough oxygen passes from your lungs into your blood, or when your lungs cannot properly remove carbon dioxide (respiratory failure)
- A skin disorder that's considered to be an allergic reaction to medicine or an infection. Symptoms may include symmetrical, red, raised skin areas that can appear all over the body, more noticeable on the fingers and toes. These patches often look like "targets" (dark circles with purple-grey centers) (erythema multiforme)
- Abnormally excessive sweating involving the arms, legs, hands and feet, underarms, and face, usually unrelated to body temperature or exercise
- Blistering of the skin or mouth caused by the immune system attacking healthy tissue (pemphigoid)
- Decreased secretion of hormones produced by adrenal glands
- Decreased thyroid stimulating hormone: a lab test result associated with abnormal thyroid function
- Dehydration
- Dry eye
- Flu like symptoms (which may include fever, chills, cough, sore throat, runny or stuffy nose, muscle or body aches, headaches, feeling tired)
- Hair loss
- Heart rate increased
- Heart rhythm abnormal
- Hives

Steven Park, MD


- Inflammation of the eye
- Inflammation of the kidney
- Inflammation of the lining of bronchial tubes, which carry air to and from the lungs (bronchitis)
- Inflammation of the liver
- Inflammation of the muscle
- Inflammation of the pancreas
- Inflammation of the pituitary gland
- Inflammation of the stomach
- Inflammation of the thyroid gland
- Joint pain or stiffness
- Kidney function failure, kidney disease
- Low blood pressure
- Low white blood cell counts (neutropenia): these put you at higher risk for infection
- Skin disease with thickened patches of red skin, often silvery scales (psoriasis)
- Trouble falling and/or staying asleep (insomnia)
- Underactive function of the pituitary gland situated at the base of the brain
- Vision blurred

Rare side effects of nivolumab include [greater than or equal to 1/10,000 to less than 1/1,000 or greater than or equal to 0.01% to less than 0.1%]:

- A disease involving abnormal collections of inflammatory cells (granulomas) in organs such as lungs, skin, and lymph nodes (sarcoidosis)
- A disease that may affect your body's defense system, called immune system. Certain white blood cells may attack other blood cells. These abnormal blood cells collect in your spleen and liver, causing these organs to enlarge. The symptoms may include fever, rash, and low blood cell counts (hemophagocytic lymphohistiocytosis (HLH) syndrome)
- A malfunction of the immune system that produces autoantibodies, which attack red blood cells as if they were foreign substances to the body (autoimmune hemolytic anemia)
- A neuromuscular disease that may cause weakness of eye, face, breathing, and swallowing muscles (myasthenic syndrome, myasthenia gravis)
- A severe skin disease characterized by blistering and peeling of the top layer of skin resembling a severe burn (toxic epidermal necrolysis) which can be serious and potentially life-threatening
- A swelling and irritation of the thin saclike membrane surrounding the heart (pericardium) (pericarditis)
- Acne-like skin condition resulting in redness of face (rosacea)
- An autoimmune disorder associated with progressive muscle weakness or paralysis (Guillain-Barre syndrome)

Steven Park, MD


- An inflammatory disorder that causes muscle pain and stiffness, especially in the shoulders (polymyalgia rheumatica)
- Cranial nerve disorder: an impairment of one of the twelve cranial nerves that can cause pain, tingling, numbness, weakness, or paralysis of the face including the eyes
- Damage to the protective covering of the nerves in the brain and spinal cord
- Diabetes complications resulting in excess blood acids
- Disease caused by the body's immune system attacking healthy organs (autoimmune disorder)
- Disorder of the lymph nodes which causes the lymph nodes to become enlarged, inflamed and painful, commonly affecting lymph nodes of the neck and possibly associated with fever or muscle and joint pains (histiocytic necrotizing lymphadenitis or Kikuchi lymphadenitis)
- Double vision
- Drug induced liver injury
- Inflammation of blood vessels
- Inflammation of the brain
- Inflammation of the heart
- Inflammation of the lining of the brain and spinal cord
- Inflammatory disorder of skin and mucous membranes, resulting in blistering and shedding of skin (Stevens Johnson syndrome) which can be serious and potentially life-threatening
- Lung infiltrates, associated with infection or inflammation
- Muscle fiber released into the blood stream which could damage your kidneys (rhabdomyolysis)
- Rupture of the intestine/hole in the intestine or stomach
- Severe allergic reaction may include but not limited to high grade fever, rash, swelling and pain

The following events have been identified during post-approval use of nivolumab. Because reports are voluntary from a population of unknown size, an estimate of frequency cannot be made. The events may be serious or life threatening.

- A condition that occurs when donor bone marrow or stem cells attack the recipient (graft-versus-host disease)
- A disease that may affect several parts of the body, including the eyes, ears, nervous system, and skin. The symptoms may include eye swelling, pain and/or blurred vision; hearing loss, ringing in the ears; and /or loss of skin color (Vogt-Koyanagi-Harada (VKH) disease)
- Solid organ transplant rejection

# Additional information on lung inflammation (pneumonitis):

The study staff will watch you closely for changes in your ability to breathe and for other signs or symptoms that might show you are developing t lung inflammation and will perform regular tests including physical exams, measurement of oxygen levels through non-invasive testing (for example, pulse oximeter), blood tests, chest x-rays and/or CT scans.

Steven Park, MD


Please inform study staff AT ONCE if you experience any of the following:

- Any new or increased shortness of breath
- Any new or increased chest pain
- Any new or increased pain/difficulty while breathing
- Any new or increased cough or any significant change in your type of cough; for Example, any new or increased mucous or blood in your cough
- Any change in the amount of oxygen you require
- Any fever, fatigue, or other symptoms that occur at the same time as any changes to your breathing or other lung symptoms

If you start to develop symptoms, your study doctor will ask you to return to the clinic for additional tests, which could include a physical exam, measurement of oxygen levels, blood tests, chest x-rays, and/or CT scans. You will be monitored very closely for changes in your overall lung symptoms, monitoring that may require hospitalization. You may require specific treatment in order to control pneumonitis. You may also be seen by a special doctor called a pulmonologist, who has special training to be an expert in how your lungs work.

Prolonged treatment with medicines that suppress inflammation, sometimes needed to manage the side effects of nivolumab study treatment, may lower your body's ability to fight off certain infections (such as opportunistic infections). These infections may require treatment with antibiotic or antifungal medications and may be fatal.

# Additional information on transplant risks:

Complications, including fatal events, have occurred in subjects who received allogeneic hematopoietic stem cell transplantation (HSCT) before or after nivolumab.

Complications, including rejection, have also been reported in subjects who have received an organ or tissue transplant. Treatment with nivolumab may increase the risk of rejection of the organ or tissue transplant.

## Blood Draw/IV/Catheter Insertion Risks

You may have pain or bruising at the site where the blood is drawn, or IV is inserted. You may feel faint. An infection at the site of the blood draw or IV insertion is possible.

#### Allergic Reaction Risks

As with taking any drug, there is a risk of allergic reaction. If you have a very serious allergic reaction, you may be at risk of death. Some symptoms of allergic reactions are:

Steven Park, MD


- Rash
- Wheezing and difficulty breathing
- Dizziness and fainting
- Swelling around the mouth, throat or eyes
- A fast pulse
- Sweating

Please seek treatment immediately and tell the study doctor and study staff if you have any of these symptoms, or any other side effects, during the study.

#### **MRI Risks**

There are very few risks known to be associated with MRI scans. The only risks relate to the presence of loose metalwork in the body (for example, surgical artery clips or foreign bodies) and subjects with pacemakers.

There are risks with an MRI if you are pregnant or have one of the following: an artificial heart valve, metal plate, pin or other metallic objects in your body (including a bullet or shrapnel). During an MRI, you will have to lie still on your back in the MRI scanner in a tight space. This may make you anxious. The MRI scan does not cause any pain and does not expose you to x-ray radiation.

#### **Lumbar Puncture Risks**

Lumbar puncture (spinal tap) is performed in the lower back, in the lumbar region. During lumbar puncture, a needle is inserted between two lumbar bones (vertebrae) to remove a sample of cerebrospinal fluid — the fluid that surrounds your brain and spinal cord to protect them from injury. Side effects include:

- Headache
- Nausea
- Vomiting dizziness
- Back pain or discomfort
- Bleeding at puncture site or rarely into epidural space

### Reproductive Risks

## Women Who Can Get Pregnant or Are Breastfeeding

You may not take part in this study if you are breastfeeding, are pregnant, think that you may be pregnant, or are trying to get pregnant. If you are pregnant or breastfeeding, there may be risks to you and the baby that are not known at this time. Women who can get pregnant will be tested for pregnancy before and during the study.

Steven Park, MD


You must avoid getting pregnant in order to take part in this research study. You should not have sexual intercourse, or you should use a highly effective contraceptive method for the duration of this study and for up to 5 months after the last dose of study drug.

You should not breastfeed while receiving the study drug and for up to 5 months from the last dose of the study drug.

It is important for you to tell the study doctor at once if you get pregnant or think that you might be pregnant while you are in the research study. If this happens, the study doctor will discuss with you what you should do. If you get pregnant, you will be asked to stop taking part in the study. You may also be asked questions about your pregnancy and the baby.

#### Unknown Risks

You might have side effects or discomforts that are not listed in this form. Some side effects may not be known yet. New ones could happen to you. Tell the study doctor or study staff right away if you have any problems.

#### ALTERNATIVES TO BEING IN THE STUDY

You do not need to take part in this research study. You may choose not to take part in this study and receive other available treatments for primary CNS lymphoma as recommended by your study doctor, such as standard chemotherapy, standard radiation therapy, steroid therapy, other medications, or you may be eligible for other experimental treatments for primary CNS lymphoma.

As an alternative to taking part in this study, you may receive treatment to just control the symptoms you are having because of your disease. You can also choose to have no treatment at all. Your study doctor can discuss the alternatives and the risks and benefits of these alternatives with you.

# POTENTIAL BENEFITS OF BEING IN THE STUDY

Taking part in this study may or may not improve the symptoms of your condition. There may be no benefit to you and your condition may not improve. While you are in this study, your study doctor will follow your condition closely. By taking part in the study you may help people in the future.

#### **COSTS OF BEING IN THE STUDY**

You or your insurance company will be charged for routine medical care and/or hospitalization in the usual manner. You or your insurance company will not be charged for procedures that are being performed for research purposes only. The study drug (nivolumab) will be provided at no cost to you. Some health insurance plans may not cover certain procedures and medical treatments. You

Steven Park, MD


may wish to discuss coverage with your insurance company before agreeing to participate in this study.

For more information on clinical trials and insurance coverage, you can visit the National Cancer Institute's web site at <a href="http://cancer.gov/clinicaltrials/understanding/insurance-coverage">http://cancer.gov/clinicaltrials/understanding/insurance-coverage</a> You can print a copy of the "Clinical Trials and Insurance Coverage" information from this web site. Another way to get the information is to call 1-800-4-CANCER (1-800-422-6237) and ask them to send you a free copy.

#### YOUR PAYMENT FOR BEING IN THE STUDY

You will not be paid for being in this study. You will also not be paid or reimbursed for time and transportation costs for traveling to and from the clinic.

### STUDY STAFF PAYMENT/FINANCIAL DISCLOSURE

None of the doctors asking you to participate in this study has received or will receive money or other benefits for personal use from the company (BMS) that developed the study drug, nivolumab, used in this study. However, BMS will give money or other benefits to a research fund, foundation, educational institution, or other organization with which the doctor or study staff is associated.

# **COMPENSATION FOR INJURY**

In the event that you are harmed as a result of your participation in this study, we will provide or arrange for treatment as necessary. This treatment, as well as other medical expenses, will be billed to you or your insurance company in the usual manner. You do not waive any legal rights by signing this consent form.

If you become ill or are hurt while you are in the study, get the medical care that you need right away.

Treatment for research-related injuries will be billed to you or your insurance in the usual manner. Neither the sponsor nor BMS will provide compensation for research-related injuries or the treatment of such injuries.

In no way does signing this consent form waive your legal rights nor does it relieve the investigators, Sponsor, or involved institutions from their legal and professional responsibilities.

Steven Park, MD


#### CONFIDENTIALITY

The records of this study will be kept private. If any report about this research is published, we will not include any information that will make it possible to identify you. However, there is some risk that de-identified data might be re-identified. Also, your record for this study may be reviewed and/or photocopied, by Atrium Health, or by representatives of the Food and Drug Administration or other government agencies.

To ensure that your information collected for this study will be kept private, your name will not be used whenever possible. A code will be used instead of your name. All of your study data will be kept in a secure location.

Your de-identified samples (with only your unique ID number) and associated data will be stored in a biospecimen repository (a "bank" of specimens and data) at Atrium Health.

Your samples may be used to determine the sequence of some or all of your genes (DNA – traits passed in families). However, this study is not intended to identify disease causing mutations that can affect the health of close family members (such as your parents, siblings, or children). All specimens collected for the purposes of this study will be considered donated materials and will be stored no longer than 15 years. You will not receive any results from any analyses performed on blood and/or bone marrow collected for research purposes.

# <u>AUTHORIZATION TO USE AND DISCLOSE YOUR PROTECTED HEALTH INFORMATION</u>

| If you wish to participate in this research study, you |
|--------------------------------------------------------|

Printed Name of Research Subject

must sign this Authorization. By signing this Authorization, you give all healthcare providers, including Atrium Health, permission to use or disclose (release) your protected health information, both past and present, for the research study described here:

**LCI-HEM-PCNSL-RMPV-001:** Phase 1B Trial of Nivolumab Consolidation Following Completion of Standard High Dose Methotrexate Containing Induction Chemotherapy in Older (≥ 65) Patients with Primary CNS Lymphoma

The protected health information that we may use or disclose (release) for this research may include all information in your medical record, such as results of physical examinations, medical history, lab tests, or certain health information indicating or relating to a particular condition.

Steven Park, MD


The health information listed above may be used by and/or disclosed (released) to:

- Study investigator and research staff
- Study sponsor and/or its associated companies
- Regulatory or other governmental authorities of the United States or other countries based on this study
- Other persons or agents authorized by the study sponsor (including BMS)
- Atrium Health employees
- Other persons or agencies as required by law or allowed by federal regulations
- Advarra Institutional Review Board (Advarra IRB) or Data Safety and Monitoring Boards.

Atrium Health is required by law to protect your protected health information. By signing this Authorization, you authorize Atrium Health to use and/or disclose (release) your protected health information for this research study. Those persons who receive your protected health information may not be required by Federal privacy laws (such as the Privacy Rule) to protect it and may share your protected health information with others without your permission, if permitted by laws governing them. Your protected health information may then no longer be protected by the Privacy Rule.

Please note that you do not have to sign this Authorization, but if you do not, you may not receive research-related treatment through this study. However, Atrium Health may not condition (withhold or refuse) your other Atrium Health providers treating you on whether you sign this Authorization. You may change your mind and withdraw (take back) this Authorization at any time, except to the extent that Atrium Health or the Sponsor has already used or disclosed your protected health information based on this Authorization. To withdraw this Authorization, you must write to the Study Doctor at the address listed on the first page of this form.

No publication or public presentation about the research described above will reveal your identity without another Authorization from you. If all protected health information that does or can identify you is removed, the remaining information will no longer be subject to this Authorization or federal rules (such as the Privacy Rule) and may be used or disclosed for other purposes.

When the research for which the use or disclosure is made involves treatment and is conducted by Atrium Health: To maintain the integrity of this research study, you generally will not have access to your personal health information related to this research until the study is complete.

At the conclusion of the research study and at your request, you generally will have access to your protected health information. Access to your protected health information in a medical record is described in the Notice of Privacy Practices provided to you by Atrium Health.

Steven Park, MD


When conducting research, the data and results may be used or disclosed for further treatment outcomes research or to research a secondary result. This Authorization will remain in effect after the end of the current study, and any future related secondary study unless it is revoked by the you in writing as described above.

Signature of Research Subject or Research Subject's Legally Authorized Representative

Printed name of Research Subject or Research Subject's Legally Authorized Representative

Date

# WHOM TO CONTACT ABOUT THIS STUDY

During the study, if you experience any medical problems, suffer a research-related injury, or have questions, concerns or complaints about the study, please contact the Investigator at the phone number listed on the first page of this consent document. If you seek emergency care, or hospitalization is required, alert the treating physician that you are participating in this research study.

An institutional review board (IRB) is an independent committee established to help protect the rights of research subjects. If you have any questions about your rights as a research subject, and/or concerns or complaints regarding this research study, contact:

By mail:

Advarra IRB

or call collect:

or by email:

Please reference the following number when contacting the Study Subject Adviser: <u>Pro00036735.</u>

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

Steven Park, MD


#### BEING A STUDY VOLUNTEER AND WITHDRAWING FROM THE STUDY

Your participation in this study is completely voluntary. You should feel under no pressure to be in the study. If you decide not to be in the study, that will not in any way harm your relations with your doctors or with Atrium Health. You are free to stop being in the study if you change your mind after entering it. This would not harm your relations with your doctors or Atrium Health.

If you choose to withdraw from the study, please notify the study doctor on page 1 of this consent form.

Any specimens which may have been collected but have not yet been processed may be destroyed upon your written request. No specimens will be returned to you. If you leave the study for any reason, you will be asked to have the procedures completed for the final visit.

Your part in the research may stop at any time for any reason, such as:

- The sponsor or the study doctor decides to stop the study.
- The sponsor or the study doctor decides to stop your part in the study for your safety.
- You need additional medicine.
- You do not follow the study rules.
- You have a new injury or illness.
- You decide to stop.

You may be asked to stop the study even if you do not want to stop.

## NEW INFORMATION ABOUT THE STUDY

Any new important information that is discovered during the study and which may influence your willingness to continue participation in the study will be provided to you.

Steven Park, MD


# STATEMENT OF CONSENT

| the purposes listed above | nd its contents were explain<br>we. All of my questions we<br>of this form for my record | ere answered to | my satisfaction. | I will receive a |
|---|---|---|---|---|
| Signature of Research S | pubject | | //<br>Date | Time |
| Printed Name of Resea | rch Subject | | | |
| Signature of Legally Au | thorized Representative (i | f applicable) | ////// | Time |
| Printed Name of Legall | y Authorized Representat | ive (if applicable) | ) | |
| STATEMENT OF P | ERSON EXPLAINING | CONSENT | | |
| and purpose of the abo<br>legally authorized repre | ed to the subject or the su<br>ve study. There has been<br>sentative to ask questions<br>hat the subject or the subject | an opportunity f<br>about this resear | or the subject or<br>rch study. I have<br>orized representat | the subject's<br>been available to<br>tive has about this |
| Signature of Person Ex | plaining Consent | | //<br>Date | Time |
| Printed Name of Perso | n Explaining Consent | | | |
| Steven Park, MD | Advarra IRB Approved | l Version 25 Aug 2022 | | Revised 25 Aug 2022 |
| | | Affix Part | icipant Barcode L | abel Here |